CLINICAL TRIAL: NCT06008964
Title: Determination of the Effect of Aromatherapy Using Lavender and Ylang Ylang Essential Oils on Pain Severity and Comfort Level After Cesarean Section: A Randomized Controlled Study
Brief Title: The Effect of Aromatherapy Applied After Cesarean Section on Pain Intensity and Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Şerife İrem DÖNER (Unknown); Merve YAZAR (Unknown); JULE ERİÇ HORASANLI (Unknown)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, LECTURER, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Aromatherapy Group
Record Dates: First submitted 2023-04-18; First posted 2023-08-24 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Section Complications
Keywords: Aromatherapy; pain; ceserean
MeSH Terms: conditions — Pain | interventions — Inhalation; lavender oil

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ylang Ylang oil Group (Active Comparator): GROUP 1
  Interventions: Other: Ylang Ylang oil with inhalation
- Control Group (No Intervention): No intervention
- Lavender oil (Active Comparator): GROUP 2
  Interventions: Other: Lavender oil with inhalation

INTERVENTIONS:
Other: Ylang Ylang oil with inhalation — Ylang Ylang OIL WILL BE INHALED
  Arms: Ylang Ylang oil Group
Other: Lavender oil with inhalation — LAVENDER OIL WILL BE INHALED
  Arms: Lavender oil

SUMMARY:
Today, many complementary therapies such as acupuncture, reflexology, homeopathy, hypnotherapy, music and aromatherapy are tried in addition to medical methods to reduce pain and anxiety. Aromatherapy is a therapy method in which essential oils are used to protect and improve physical and psychological health. Oils can be applied directly to a single person or indirectly to people in a room by inhalation . In direct application without steam, essential oils can be applied by inhalation by dripping onto a cotton ball . It is stated that lavender aromatherapy, one of the most commonly used aromatherapies, has analgesic, antiseptic, sedative, antispasmodic and healing properties Ylang Ylang aromatherapy is stated analgesic, anti-inflammatory, antimicrobial, antiemetic,anti-tarral, carminative, sedative, antiseptic, spasmolytic properties. In the studies conducted, anxiety, labor pain, labor duration, and psychological effects of aromatherapy were examined, but no study was found in which lavender and chamomile essential oils were used and the effects of pain and comfort level were examined. The aim of this study is to determine the effect of lavender and Ylang Ylang essential oils in relieving pain and increasing comfort after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years old,
* women who have had a cesarean section

Exclusion Criteria:

* epilepsy,
* migraine,
* chronic headache,
* asthma,
* women who are allergic to fragrance sensitivities to aromatic oils

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 18-49 who have undergone cesarean section
Enrollment: 96 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
pain related to cesarean section | post operative 4-8-12 hours
  It will be measured with Visual Analog Scale. Visual Analog Scale has a rating between 0-10. The higher the score, the greater the pain.

SECONDARY OUTCOMES:
comfort related to cesarean section | post operative 4-8-12 hours
  Comfort will be measured with the postpartum comfort scale. The higher the score, the higher the comfort level.

CONTACTS AND LOCATIONS:
Overall Officials: şerife irem döner, Study Chair — serifeiremdoner@gmail.com; Merve Yazar, Study Chair — merve.yazar@karatay.edu.tr
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No